CLINICAL TRIAL: NCT05101941
Title: Evaluating the Osseointegration of Immediate Dental Implant Placed in the Presence of Chronic Inflammatory Periapical Lesions
Brief Title: Immediate Dental Implant Placed in the Presence of Chronic Inflammatory Periapical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Immediate implants_2020
Record Dates: First submitted 2021-10-20; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Immediate Dental Implant; Tooth Exratction; Periapical; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immediate dental implants (Experimental)
  Interventions: Procedure: Immediate dental implants

INTERVENTIONS:
Procedure: Immediate dental implants — Implants will be immediately placed in sockets associated with chronic periapical granuloma Extraction of non-restorable Teeth with periapical granuloma and socket debridement will be done then implants will be placed

SUMMARY:
Compromised teeth with periapical pathologies are removed before dental implant placement and sockets are left to heal.

Some clinicians began to immediately place dental implants in fresh extraction sockets associated with chronic inflammatory periapical lesions and these studies revealed high success rates

DETAILED DESCRIPTION:
12 implants will be immediately placed in sockets associated with chronic periapical granuloma. Clinical (Wound healing, Pain, swelling, implant stability) and radiographic parameters (Peri-implant radiolucency) will be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ranging from 18 to 45 years with no gender predilection agreed to come for minimum follow-up visits for 6 months.
* Adequate bone beyond teeth apices without jeopardizing any anatomical structure.
* Single rooted mandibular teeth with chronic inflammatory periapical lesions represented as periapical radiolucency, pulp necrosis, sinus tract, failed RCT.

Exclusion Criteria:

* Smokers and alcoholics.
* Medically compromised patients having uncontrolled diabetes or coagulation disorders.
* Restorable teeth.
* Periodontitis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
Change in Implant stability | immediately, at 3 months and 6 months
  It will be measured by implant stability meter (Osstell™)
Change in peri implant radiolucency | immediately, and 6 months
  Immediate post-operative and after 6 months CBCT will be requested in order to compare the dimension of the periapical lesion in millimeters using OnDemand system.

SECONDARY OUTCOMES:
Change in pain score | within a week
  It will be recorded daily for the first week through a 10-point Visual Analogue Scale (VAS) from 0 to 10 (0-1= None, 2-4= Mild, 5-7= Moderate, 8-10= Severe).
Change in swelling status | within a week
  It will be recorded daily for the first week through a 10-point scale with 4 parameters will be used.
  none (no swelling), light (intraoral, localized to the treated area), moderate (extraoral swelling localized to the treated area), and severe (extraoral swelling extending beyond the treated area)
Change in Early Wound Healing Index | at 2 weeks, 4 weeks, and 8 weeks
  Using Early Wound Healing Index (EHI), it will be evaluated across weeks 2, 4 and 8.
  (EHI; 1: complete flap closure-no fibrin line; 2: complete flap closure-fine fibrin line; 3: complete flap closure-fibrin clot; 4: incomplete flap closure-partial necrosis; 5: incomplete flap closure-complete necrosis).

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt